CLINICAL TRIAL: NCT00654732
Title: A Randomized Phase II Study of Rituximab With ABVD Versus Standard ABVD for Patients With Advanced-Stage Classical Hodgkin Lymphoma With Poor Risk Features (IPS Score > 2)
Brief Title: Combination Chemotherapy With or Without Rituximab in Treating Participants With Stage III-IV Classic Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0144; NCI-2018-01855 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2007-0144 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Classic Hodgkin Lymphoma; Lugano Classification Stage III Hodgkin Lymphoma AJCC v8; Lugano Classification Stage IV Hodgkin Lymphoma AJCC v8
MeSH Terms: interventions — Bleomycin; Dacarbazine; Doxorubicin; Rituximab; CT-P10; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (rituximab, combination chemotherapy) (Experimental): Participants receive rituximab intravenously IV over 7 hours on days 1, 8, 15, and 22 of course 1 and on days 1 and 8 of course 2. Participants also receive doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine IV over 1 hour on days 1 and 15. Treatment with ABVD repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bleomycin; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Biological: Rituximab; Drug: Vinblastine
- Arm B (combination chemotherapy) (Active Comparator): Participants receive doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine as in Arm A.
  Interventions: Drug: Bleomycin; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Drug: Vinblastine

INTERVENTIONS:
Drug: Bleomycin — Given IV
  Other Names: BLEO; BLM
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
  Arms: Arm A (rituximab, combination chemotherapy)
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; VLB

SUMMARY:
This phase II trial studies how well combination chemotherapy with or without rituximab works in treating participants with stage III-IV classic Hodgkin lymphoma. Monoclonal antibodies, such as rituximab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving rituximab with combination chemotherapy may work better in treating participants with classic Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the event free survival (EFS) following therapy with rituximab plus adriamycin (doxorubicin hydrochloride), bleomycin, vinblastine, and dacarbazine (ABVD) or standard ABVD in patients with newly diagnosed classical Hodgkin lymphoma who have poor prognosis defined as International prognostic score (IPS) of > 2.

SECONDARY OBJECTIVES:

I. To compare the effect of the two treatment arms on positron emission tomography (PET) scan results after 2 cycles of therapy.

II. To compare the effect of the two treatment arms on the level of circulating malignant Hodgkin stem cells.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Participants receive rituximab intravenously (IV) over 7 hours on days 1, 8, 15, and 22 of course 1 and on days 1 and 8 of course 2. Participants also receive doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine IV over 1 hour on days 1 and 15. Treatment with ABVD repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Participants receive doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine as in Arm A.

After completion of study treatment, participants are followed up every 3 months for the first year, every 4 months for the second year, every 6 months for years 3-5, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patient with classical Hodgkin's lymphoma patients with stage III and IV
* International Prognostic Score of > 2 (patient must have > 2 of the following risk features: Male, >= 45 years of age, stage IV, albumin < 4, white blood cell count [WBC] >= 15, lymphocytes < 8% or < 600, hemoglobin [Hgb] < 10.5)
* Must sign a consent form
* Absolute neutrophil count (ANC) >= 1,500/microL
* Platelet > 100,000/microL
* Left ventricular ejection fraction (LVEF) >= 50% by multigated acquisition (MUGA) scan or echocardiogram
* Serum creatinine < 2 mg/dl
* Serum bilirubin < 2 mg/dl
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2 x upper limit of normal (ULN)
* Bi-dimensionally measurable disease

Exclusion Criteria:

* Lymphocyte predominant Hodgkin's lymphoma
* Known human immunodeficiency virus (HIV) infection
* Pregnant women and women of child bearing age who are not practicing adequate contraception
* Prior chemotherapy or radiation therapy
* Severe pulmonary disease as judged by the principal investigator (PI) including chronic obstructive pulmonary disease (COPD) and asthma
* Active infection requiring treatment with intravenous therapy
* Presence of central nervous system (CNS) lymphoma
* Concomitant malignancies or previous malignancies within the last 5 years (exception made for adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of cervix)
* Active hepatitis B or C infection

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-03-19 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hun Lee, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Frontline advance stage hodgkin lymphoma
Groups:
- RABVD: Rituximab Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine
- ABVD: Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine
Period: Overall Study
Arm/Group | RABVD | ABVD
Started | 26 | 32
Completed | 22 | 26
Not Completed | 4 | 6
Not completed — Adverse Event | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RABVD | ABVD | Total
Number analyzed (Participants) | 26 | 32 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 11 | 16 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 14 | 22 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — The study did not discriminate against race/ethnicity. | NA — The study did not discriminate against race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — The study did not discriminate against race/ethnicity. | NA — The study did not discriminate against race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — The study did not discriminate against race/ethnicity. | NA — The study did not discriminate against race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — The study did not discriminate against race/ethnicity. | NA — The study did not discriminate against race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — The study did not discriminate against race/ethnicity. | NA — The study did not discriminate against race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — The study did not discriminate against race/ethnicity. | NA — The study did not discriminate against race/ethnicity. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 26 | 32 | 58
Region of Enrollment [Number; unit: participants]
  United States | NA — This information was not collected | NA — This information was not collected | NA — This information was not collected

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Rate
Description: EFS will be estimated using the Kaplan-Meier method. The log-rank test will be performed to test the difference in time-to-event distributions between patient groups. Cox proportional hazards model will be utilized to include multiple covariates in the time-to-event analysis. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate.
Time Frame: From the start of study treatment up to 3 years
Measure: Count of Participants; unit: Participants
Groups:
- RABVD: Experimental Arm Rituximab, Adriamycin, Bleomycin, Vinblastine, and Dacarbazine
- ABVD: Control Arm (Adriamycin, Bleomycin, Vinblastine, and Dacarbazine)
Arm/Group | RABVD | ABVD
Number analyzed (Participants) | 22 | 26
Participants | 17 | 20

ADVERSE EVENTS:
Time Frame: 4 years and 6 months
Groups:
- RABVD: Rituximab chemotherapy
- ABVD: Chemotherapy only
Arm/Group | RABVD | ABVD
All-Cause Mortality (participants affected / at risk) | 5/26 | 6/32
Serious Adverse Events (participants affected / at risk) | 13/26 | 13/32
Other Adverse Events (participants affected / at risk) | 0/26 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RABVD (N=26) | ABVD (N=32)
Neutropennia (Blood and lymphatic system disorders) | 13 | 13
Anemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Infection (Immune system disorders) | 4 | 1
Respiratory Complicaton (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Neuropathy (Nervous system disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT00654732/Prot_SAP_000.pdf